CLINICAL TRIAL: NCT05069324
Title: The PrOMISE Study: PegvisOMant and the Immune SystEm
Brief Title: PegvisOMant and the Immune SystEm (PROMISE)
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea M. Isidori, Full Professor, University of Roma La Sapienza
Other Study IDs: PROMISE
Record Dates: First submitted 2020-10-19; First posted 2021-10-06 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Acromegaly
Keywords: Acromegaly; Pegvisomant; Immunity; Immune function; Metabolism; Body composition; Quality of life; Sleep disturbances
MeSH Terms: conditions — Acromegaly; Parasomnias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Acromegaly patients not adequately controlled by any kind of SSAs monotherapy: Acromegaly patients not adequately controlled by any kind of SSAs monotherapy, requiring PEG in combination with SSAs or PEG monotherapy
- Acromegaly patients adequately controlled by medical treatment: Acromegaly patients adequately controlled by medical treatment, by any kind of SSAs or by PEG
- Healthy controls: Healthy volunteers matched with patients for age and sex

SUMMARY:
This is a prospective observational pilot study for the evaluation of immune cells phenotype in acromegalic patients in comparison with a control population and to investigate the impact of disease control and different medical treatments (particularly Pegvisomant) on immune function and its implication on insulin resistance, metabolic complications and fat accumulation.

DETAILED DESCRIPTION:
The observational study will concern the collection of data from patients who, as they are not controlled by SSAs therapy (cohort 1), require PEG therapy in monotherapy (group 1) or in combination with SSAs (group 2), according to common clinical practice. The investigators will enroll also acromegalic patients adequately controlled by medical therapy (cohort 2), respectively treated by any kind of SSAs (group 3) and by PEG (group 4) for comparison between different medical treatments. The data will be prospectively collected at baseline and after 8 weeks of treatment.

A control group will be enrolled including healthy volunteers matched with patients for age and sex.

The primary outcome will be the immune profiling by quantification of peripheral blood mononuclear cells (PBMC) subpopulations.

Secondary outcome measures will be

* Evaluation of inflammatory cytokines and adipokines production.
* Evaluation of glucose, insulin, c-peptide, HbA1c, triglycerides, total cholesterol, HDL-cholesterol, LDL-cholesterol apolipoprotein B and A. Insulin resistance and β cell function will be assessed by the homeostasis model assessment for insulin resistance (HOMA-IR) index and for β cell secretion (HOMA-β). Anthropometric measurements will include body weight, height and waist and hip circumference.
* Evaluation of body composition. Composite outcome measure consisting of lean mass, skeletal muscle and fat distribution analysis.
* Fasting samples from all patients will be assayed for disease control parameters.
* Evaluation of quality of life. Quality of life will be measured by Short Form (SF)-36-Item Health Survey total score, SF-36-Item Health Survey physical component summary score and SF-36-Item Health Survey mental component summary score and Acromegaly quality of life (AcroQol) questionnaire.
* Evaluation of sleep disturbances. Sleep disturbances will be measured by Epworth Sleepiness Scale (ESS) and by polysomnography when appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed acromegaly not adequately controlled by surgery and/or radiation therapy and in whom an appropriate medical treatment with any kind of somatostatin analogs (SSAs) did not control the disease or was not tolerated;
* Previously diagnosed acromegaly adequately controlled by medical treatment;
* Signed informed consent to participate in the study.

Exclusion Criteria:

* Adequately controlled disease by surgery and/or radiation;
* Patients with transaminases more than 3 times the upper limit of normal;
* Hypersensitivity to PEG or any of its ingredients;
* History of other neoplasms, radiotherapy or chemotherapy in the last 5 years;
* Clinical or laboratory signs of significant hepatobiliary, or pancreatic disease;
* Severe infections, surgery, trauma requiring hospitalization within 3 months before enrolment;
* Severe chronic kidney disease (stage 4-5);
* Any active blood or rheumatic disorders in the last 5 years;
* Pregnant or nursing women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10 patients with acromegaly not well controlled by SSAs therapy (cohort 1), requiring add PEG to SSAs or switch to PEG monotherapy, according to common clinical practice.
  20 patients adequately controlled by medical therapy (cohort 2), treated by any kind of SSAs or by PEG .
  30 age- and sex matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Peripheral blood mononuclear cell subpopulations | baseline
  Number of cells (number per mm3) of peripheral blood mononuclear cell subpopulations
Change of peripheral blood mononuclear cell subpopulations | baseline and after 8 weeks
  Number of cells (number per mm3) of peripheral blood mononuclear cell subpopulations

SECONDARY OUTCOMES:
Tumor necrosis factor alfa (TNFα) | baseline and post 8 weeks
  Chemiluminescence measurement of TNFα serum concentrations (pg/ml)
Transforming growth factor beta (TGF-β) | baseline and post 8 weeks
  Chemiluminescence measurement of TGF-β serum concentrations (pg/ml)
Interleukin-1 (IL-1) | baseline and post 8 weeks
  Chemiluminescence measurement of IL-1 serum concentrations (pg/ml)
Interleukin-6 (IL-6) | baseline and post 8 weeks
  Chemiluminescence measurement of IL-6 serum concentrations (pg/ml)
Interleukin-10 (IL-10) | baseline and post 8 weeks
  Chemiluminescence measurement of IL-10 serum concentrations (pg/ml)
Interferon gamma | baseline and post 8 weeks
  Chemiluminescence measurement of interferon gamma serum concentrations (pg/ml)
Monocyte chemoattractant protein (MCP-1) | baseline and post 8 weeks
  Chemiluminescence measurement of MCP-1 (pg/ml)
Adipokines production (visfatin) | baseline and post 8 weeks
  Measurement of visfatin serum concentrations
Adipokines production (adiponectin) | baseline and post 8 weeks
  Measurement of adiponectin serum concentrations
Adipokines production (vaspin) | baseline and post 8 weeks
  Measurement of vaspin serum concentrations
Adipokines production (omentin) | baseline and post 8 weeks
  Measurement of omentin serum concentrations
Metabolic parameters: glycemia | baseline and post 8 weeks
  Evaluation of glucose (mmol/l)
Insulin production | baseline and post 8 weeks
  Evaluation of insulin (mU/L)
Insulin secretion | baseline and post 8 weeks
  Evaluation of c-peptide (ng/ml)
Metabolic parameters: glycosylated haemoglobin | baseline and post 8 weeks
  Evaluation of HbA1c (mmol/mol)
Lipid profile: triglycerides | baseline and post 8 weeks
  Evaluation of triglycerides (mmol/l)
Lipid profile: cholesterol | baseline and post 8 weeks
  Evaluation of total cholesterol (mmol/l)
Lipid profile: HDL-cholesterol | baseline and post 8 weeks
  Evaluation of HDL-cholesterol (mmol/l)
Lipid profile: LDL-cholesterol | baseline and post 8 weeks
  Evaluation of LDL-cholesterol (mmol/l)
Lipid profile: Apo B | baseline and post 8 weeks
  Evaluation of apolipoprotein B (mmol/l)
Lipid profile: Apo A | baseline and post 8 weeks
  Evaluation of apolipoprotein A (mmol/l)
Insulin resistance | baseline and post 8 weeks
  Evaluation of the homeostasis model assessment for insulin resistance (HOMA-IR) index
beta cell function | baseline and post 8 weeks
  Evaluation of the homeostasis model assessment for β cell secretion (HOMA-β)
Body mass index (BMI) | baseline and post 8 weeks
  Body weight and height weight will be combined to report BMI in kg/m^2
Anthropometric parameters | baseline and post 8 weeks
  Waist and hip circumference will be combined to report waist-hip ratio
Body composition: lean mass | baseline and post 8 weeks
  Lean mass distribution (%) evaluated by a whole-body dual-energy x-ray absorptiometry (DEXA) scan
Body composition: fat mass | baseline and post 8 weeks
  Fat mass distribution (%) evaluated by a whole-body dual-energy x-ray absorptiometry (DEXA) scan
Biochemical control | baseline and post 8 weeks
  Fasting samples from all patients will be assayed for disease control parameters (insulin-growth factor and growth hormone)
Quality of life SF-36-Item Health Survey questionnaire | baseline and post 8 weeks
  Quality of life will be evaluated by the Physical Component score and the Mental Component score of the self administered questionnaire SF-36-Item Health Survey questionnaire.
  This questionnaire measures eight scales: physical functioning, role physical, bodily pain, general health (physical component) and vitality, social functioning, role emotional, mental health (mental component).
  Interpretation of the score will be the following: at each item of the questionnaire corresponds a percentage value (from 0% to 100%). The average of the single items constitutes the scale total percentage (from 0% to 100%); missing data are not considered during calculation. High score defines a more favorable health state
Acromegaly Quality of Life Questionnaire | baseline and post 8 weeks
  Evaluation of quality of life by the Acromegaly Quality of Life Questionnaire (ACROQOL), a disease specific questionnaire to measure quality of life in patients with acromegaly. It contains 22 items divided in two scales that measure physical and psychological aspects. Each of the 22 items of the AcroQoL is answered in a 1 to 5. A global score is obtained adding the results of the 22 items using a specific formula, from a minimum of 22 - worse QoL - until 110 - best QoL -
Sleep apnea | baseline and post 8 weeks
  Sleep disturbances will be measured by Epworth Sleepiness Scale (ESS). The ESS consists of eight questions regarding eight activities. Each of the activities listed has an assigned score from 0 to 3 that indicates how likely a person is to fall asleep during the activity:
  0 = would never doze, 1 = slight chance of dozing, 2 = moderate chance of dozing, 3 = high chance of dozing.
  The total score can range from 0 to 24. A higher score is associated with increased sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea M Isidori, PHD, Principal Investigator — Department of Experimental Medicine, "Sapienza" University of Rome
Locations (1):
- Department of Experimental Medicine, "Sapienza" University of Rome, Rome, Italy